CLINICAL TRIAL: NCT06663189
Title: Disease Modifying Therapies Withdrawal in Inactive Relapsing-remitting Multiple Sclerosis Patients Aged 55 and Over: A Multicentric, Randomized, Controlled, Open-label Clinical Trial (TWINS : Therapies Withdrawal IN Relapsing Multiple Sclerosis)
Brief Title: Disease Modifying Therapies Withdrawal in Inactive Relapsing-remitting Multiple Sclerosis Patients Aged 55 and Over (TWINS : Therapies Withdrawal IN Relapsing Multiple Sclerosis)
Acronym: TWINS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8670; 2024-513475-41-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-22; First posted 2024-10-29 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Relapsing-remitting Multiple Sclerosis (RRMS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Treatment withdrawal; patients will stop their Disease Modifying Treatment (DMT)
  Interventions: Drug: treatment withdrawal; Other: MRI; Behavioral: Quality of Life questionnaires; Other: Disability evaluation tests
- Control arm (Active Comparator): Patients will continue their DMT as per routine pratice
  Interventions: Drug: Usual DMT continuation; Other: MRI; Behavioral: Quality of Life questionnaires; Other: Disability evaluation tests

INTERVENTIONS:
Drug: treatment withdrawal — Patients will STOP their DMT
  Arms: Experimental
Drug: Usual DMT continuation — Patients will continue their DMT during the trial as usual : Interferon-β (IFN-β), glatiramer acetate, dimethyl fumarate, teriflunomide or diroximel fumarate
  Arms: Control arm
Other: MRI — Cerebral+spinal cord enhanced MRI (M0) Cerebral enhanced MRI (M6, Relapse early visit) Unenhanced cerebral MRI (M12, M18, M24, Relapse distant visit
Behavioral: Quality of Life questionnaires — EQ-5D5L: EuroQol-5-Dimension 5 levels Burden of Treatment Questionnaire (BTQ self-administered questionnaires) Hospital Anxiety and Depression (HAD) questionnaire
Other: Disability evaluation tests — EDSS: Expanded Disability Status Scale 25Foot/Walk 9-HPT:Nine Hole Peg Test

SUMMARY:
Multiple sclerosis (MS) is a chronic disease of the central nervous system (CNS) characterized by loss of motor and sensory function, that results from immune-mediated inflammation, demyelination and subsequent axonal damage. It is the most common cause of neurological disability in young adults, involving a long-term therapeutic follow-up. 85% of the patients are diagnosed with Relapsing-Remitting form of MS (RRMS). This form is characterized by clearly defined acute or subacute neurological symptoms (relapses) followed by periods of partial to complete recovery.

Disease-modifying therapies (DMT) used to treat RRMS are immunomodulatory or suppressor molecules which have proven efficacy in limiting disease activity (decreasing relapse rate and delaying time to disease progression).

However, the long-term safety of DMT is uncertain, as there is an increased risk of developing adverse events or infections (sometimes severe) such as observed in the last pandemic of COVID-19 (higher risk of infection), highlighting the need to reassess the benefit/risk ratio of maintaining immunomodulatory or suppressive therapy in the MS population. In elderly patients with comorbidity, this risk is further increased. To date, few studies on the discontinuation of treatment in elderly RRMS patients have been conducted. However, those available demonstrate that there was no difference in relapse rates between patients who continued or discontinued treatment. These results are consistent with immunosenescence studies in RRMS that suggested a negative correlation between relapse rate/inflammatory processes and age. On the contrary, there is evidence indicating a positive correlation between age and the number of infections.

In addition, in the current context in France, it is important to take into account the medico-social cost associated with long-term treatments. In France, the average estimated annual cost per patient is 12,000€, more than half of which is attributed to medications.Furthermore, with age progression, an inversion of the benefit/cost assessment has been observed in treated patients.

Considering these medical and medico-social factors, it is reasonable to question the value of continuing treatment in stable patients with RRMS over 55 years.

This is a randomized, controlled, multicentric, open-label, parallel groups, 1:1 ratio non-inferiority clinical trial, comparing (1) a group that will stop treatment, to (2) a group that will continue treatment, over the course of 2 years, to determine the survival rate without MS activity defined clinically or by imaging.

The patients in both arms will be followed over 2 years after randomization. 5 visits will be performed for all patients: inclusion/randomization visit (M0) and 4 follow-up visits every 6 months (M6, M12, M18, and M24). An additional phone call at M3 is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (male or female) aged 55 and over
2. RRMS diagnosis according to revised McDonald 2017 criteria
3. First MS symptom >5 years ago. If the date is unknown, RRMS diagnosis >5 years ago
4. Stable disease in the last 5 years according to the revised Lublin and Reingold classification characterized by :

   Stable T2 lesions documented by MRI performed at least 5 years prior to inclusion versus MRI performed within 6 months prior to the inclusion visit, AND Stable EDSS documented at least 5 years prior to inclusion versus EDSS documented within 6 months prior to inclusion visit, according to the investigator's judgment, AND The absence of relapses within 5 years prior to the inclusion visit
5. Treated with a Moderate Efficacy Therapy (MET) for at least 5 consecutive years (IFN-β, glatiramer acetate, dimethyl fumarate, teriflunomide, diroximel fumarate); switching from one first-line treatment to another is accepted if the reason for the change is related to personal convenience or intolerance to the first treatment.
6. Patient with affiliation to a social security regimen
7. Patient able to understand the objectives and risks associated with the research and to give informed consent to the study
8. Patient willing and able to comply with study procedures for the duration of the study

Exclusion Criteria:

1. Primary progressive or secondary progressive with or without relapse as defined by the revised Lublin and Reingold classification
2. Previous or ongoing treatment with a High Efficacy therapy (HET), with the exception of induction therapy (mitoxantrone, stem cell transplantation, alemtuzumab) provided that the last administration took place at least 10 years prior to inclusion.
3. Contraindication to MRI (claustrophobia, weight ≥ 140 kg, pacemaker, cochlear implants, foreign body in eye, intracranial vascular clips, surgery in the 6 weeks prior to the beginning of the study, coronary stent implanted in the 8 weeks prior to the beginning of the study,…).

   NB : Gadolinium contraindication will not prevent recruitment of the patient; in this case MRI will be carried out without contrast product injection
4. History of neurological disease affecting the central nervous system: hereditary degenerative CNS disease, degenerative cognitive disease, systemic autoimmune disease, sarcoidosis, Lyme disease…
5. Chronic disease which requires chronic treatment with corticoids or immunosuppressors
6. Uncontrolled cardiac, renal or hepatic disease
7. Patient participating in another interventional trial (drug or a medical device) or patient who are still within an exclusion period
8. Patient wishing to discontinue background therapy, whether or not they are experiencing adverse effects.
9. Patient not considering discontinuing background therapy, whether or not they are experiencing adverse effects.
10. Pregnant or breastfeeding woman
11. Patient with difficulty to read or understand French,
12. Patient subject to a legal protection measure

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Time to first clinical and/or radiological disease activity during a period of 2 years. | From enrollment to the end of study visit at 24 months
  A clinical activity (relapse) is defined by the occurrence of new or worsening of neurological symptoms linked to MS. Relapses must meet the following criteria:
  * Symptoms must last at least 24 hours, without other clinical factors leading to confusion (fever, infection, lesion, drug adverse events)
  * Must be followed by improvement or resolution of the neurological state within 30 days
  * New symptoms or worsening of neurological state must be accompanied by an objective neurologic state aggravation
  * The neurological symptom must be linked to the modified FSS (pyramidal, cerebellar, brainstem, sphincter, mental, sensory or visual functions)
  A radiological activity is defined if MRI shows either:
  * at least 3 new or enlarged T2 ≥ 3 mm on the same exam or
  * at least 3 cumulative new or enlarged T2 lesions ≥ 3 mm during follow up or
  * one enhanced gadolinium lesion compared to the previous MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas COLLONGUES, MD, PhD, Principal Investigator — University Hospital, Strasbourg, France
Locations (22):
- France (22):
  - CHU de Bordeaux-Hôpital Pellegrin, Bordeaux
  - CHU de Caen-Hôpital Côte de Nacre, Caen
  - CHU de Clermont-Ferrand-Hôpital Gabriel Montpied, Clermont-Ferrand
  - Assistance Publique des Hôpitaux de Paris (APHP)-Hôpital Henri Mondor, Créteil
  - CHU de Dijon-Hôpital du Bocage, Dijon
  - CH de Gonesse, Gonesse
  - CHU de Grenoble Alpes, La Tronche
  - Groupement des Hôpitaux de l'Institut Catholique de Lille Hôpital Saint Vincent de Paul, Lille
  - CHU de Lille-Hôpital Roger Salengro, Lille
  - CHU de Limoges-Hôpital Dupuytren, Limoges
  - Assistance Publique des Hôpitaux de Marseille (APHM)-Hôpital La Timone Adultes, Marseille
  - CHU de Montpellier-Hôpital G. De Chauliac, Montpellier
  - CHU de Nancy -Hôpital Central, Nancy
  - CHU de Nice-Hôpital Pasteur, Nice
  - CHU de Nîmes, Nîmes
  - Assistance Publique des Hôpitaux de Paris (APHP)-Hôpital Pitié-Salpêtrière, Paris
  - Fondation Ophtalmologique Rothschild, Paris
  - CHU de Rennes-C.H.R. Pontchaillou, Rennes
  - CHU de Rouen-Hôpital Charles Nicolle, Rouen
  - CHU Nantes -CIC de Neurologie, Saint-Herblain
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU de Tours, Tours